CLINICAL TRIAL: NCT05836467
Title: Is Myocardial Revascularization Really Necessary in Patients With ≥50-70% Coronary Stenosis Undergoing Valvular Surgery?
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: NO-CABG
Record Dates: First submitted 2023-01-27; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Heart Valve Diseases
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Valvular interventions — Any kind of intervention on heart valves

SUMMARY:
It is well documented in the literature that myocardial revascularization during valve surgery increases the risk of early mortality and morbidity.

According to the most recent version of the European Guidelines, the possibility of myocardial revascularization via coronary artery bypass should be evaluated in patients with an indication for surgical treatment of heart valve disease but with coronary artery stenosis ≥ 50-70%.

In this study, patients hospitalized for surgical heart valve disease, with occasional pre-operative finding of ≥ 50-70% coronary artery stenosis, without angina, are examined. After interdisciplinary discussion in the Heart Team, it was decided not to treat coronary artery disease during valve surgery. The aim is to evaluate the short and medium-term results of this "conscious omission".

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* Presence of valve disease of surgical interest.
* Occasional pre-operative finding of coronary stenosis >= 50-70%.

Exclusion Criteria:

* angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any valvulopathy requiring sugery, with also critical coronary stenosis of 50-70% or more.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Survival | through study completion, a minimum of 18 months
Percutaneous revascularization risk | through study completion, a minimum of 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele - Cardiac Surgery Department, Milan, Italy

IPD SHARING:
Plan to Share IPD: No